CLINICAL TRIAL: NCT05825690
Title: Investigating the Prognostic Role of Brain MRI in Anti-LGI1 Encephalitis
Brief Title: BRIEF TITLE * (in English and Sufficiently Descriptive) Role of MRI in Anti-LGI1 Encephalitis
Acronym: LGI1-IRM
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 22-5017
Record Dates: First submitted 2023-02-14; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Autoimmune Encephalitis
Keywords: Autoimmune encephalitis; LGI1 antibodies; MRI
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LGI1- Patients: Patients affected by autoimmune encephalitis with antibodies against LGI1
  Interventions: Other: Retrospective evaluation of specific brain MRI features

INTERVENTIONS:
Other: Retrospective evaluation of specific brain MRI features — Initial brain MRI and subsequent follow-up studies will be reviewed to document the presence of specific MRI features, and their association with greater disease severity in the acute phase and/or neurological sequelae after encephalitis resolution will be investigated. More specifically, we will analyze the presence of:
  * Brain MRI changes in the acute stage, i.e. < 3 months from symptoms onset, including abnormal signal intensity, altered diffusion and/or contrast enhancement in the hippocampus (unilateral/bilateral), abnormal signal intensity in basal ganglia, insula, and/or perisylvian cortex, presence of global brain atrophy, presence of hippocampal atrophy and/or MTS, hippocampal volumetry
  * Brain MRI changes after acute phase resolution (> 6 months after symptoms onset) including abnormal signal intensity in the hippocampus (unilateral/bilateral), presence of global brain atrophy, presence of hippocampal atrophy and/or MTS, hippocampal volumetry

SUMMARY:
The term "autoimmune encephalitis" denotes an heterogenous group of diseases commonly associated with autoantibodies targeting neural or glial antigens. Patients harboring antibodies against the leucine-rich glioma-inactivated protein 1 (LGI1) usually respond well to immunotherapy, but a significant percentage develop cognitive sequelae and disability nonetheless. These patients would likely benefit for more aggressive and prolonged immunotherapy, aiming to prevent permanent neurological deficits. Identifying features predicting poor outcome would be crucial to guide treatment decisions. Brain magnetic resonance imaging is a key diagnostic tool in the acute phase, but radiological changes may also appear in follow-up studies, including global brain atrophy, hippocampal atrophy and mesial temporal sclerosis. We hypothesize that specific changes identifiable in the acute and chronic phase underlie a higher risk of poor outcome and persistent neurological deficits.

ELIGIBILITY:
Inclusion Criteria:

* - Patients with a definite diagnosis of LGI1-antibody-associated encephalitis
* available MRI records
* Ascertained positivity for LGI1-antibodies in serum and/or CSF

Exclusion Criteria:

* - Positivity for another antibody against neural or glial antigens
* MRI images not available
* Not enough clinical data to ascertain outcome

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be included from the from the database of the French Reference Centre for Paraneoplastic Neurological Syndromes and Autoimmune Encephalitis (Lyon, France)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Cognitive dysfunction and disability | 12 months
  Main outcome measures will include cognitive dysfunction measured by appropriate neuropsychological evaluations, and psychiatric symptoms; it will be "none", "light", "moderate", "severe"

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites autoimmunes, Lyon, France